CLINICAL TRIAL: NCT03080389
Title: Are Extended Urine Cultures More Sensitive Than Standard Urine Cultures in Diagnosing Urinary Tract Infections in Patients With Urgency and Frequency?
Brief Title: Sensitivity of Extended Cultures in Diagnosing Urinary Tract Infections
Status: Terminated | Type: Observational
Why Stopped: Study staff not available to complete the trial
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Eric Hurtado, Urogynecology Staff, The Cleveland Clinic
Other Study IDs: FLA 16-108
Record Dates: First submitted 2016-12-20; First posted 2017-03-15 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Overactive Bladder; Overactive Detrusor; Urgency-Frequency Syndrome; UTI
Keywords: overactive bladder; overactive detrusor; urgency-frequency; urinary tract infection
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine specimens will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Extended urine culture: Each patient will be their own control and two specimens will be obtained from each participant. The first will be a catheterized urine sample to be sent for routine culture and the second will be collected from the same catheterized specimen and sent for extended culture.
  Interventions: Procedure: Extended Urine Culture

INTERVENTIONS:
Procedure: Extended Urine Culture — Extended Urine Culture Standard cultures will include 0.001 ml of specimen plated on sheep blood agar and MacConkey agar. Plates were inoculated and incubated at 35 degrees Celsius for 24 hours. Samples were considered positive if there were 10^3 cfu or greater. The extended urine culture will be spun down by centrifuge (3000 rpm for 5 min) and 0.1 ml of the sediment will be cultured for 48 hours.
  The participants will fill out the Bother, UDI-6, and PUF questionnaires before the cultures. If a patient has a positive urine culture, the patient will be asked to repeat the questionnaires 7-30 days post treatment with antibiotics. A comparison will be made between the standard and extended urine cultures to assess for a difference in identification and treatment of uropathogens.

SUMMARY:
There is some evidence to suggest standard urine cultures may not be adequate in identifying patients with low grade urinary tract infections. Therefore, there are patients with symptoms of frequency and urgency, being misdiagnosed with overactive bladder due to negative urine cultures. If this is true, could extended cultures be used to identify the false negative patients?

DETAILED DESCRIPTION:
In 2014, Hilt, Evann et al published a study called "Urine is not sterile," in which it was found via PCR and extended urine cultures, there is a microbiome that exists within the urinary bladder. In this study, 92% of the bacteria failed to be identified by a standard urine culture but 80% were identified with extended urine cultures. In further explorations of the significance of this microbiome, Pearce, Meghan et al. found that the female bladder consists of increased abundance of bacteria in patients with UUI; including Gardnerella and Lactobacilus gasseri. Then in 2015, a study by Thomas-White, Krystal et al. found that patients with urge urinary incontinence (UUI) who responded to treatment with Solifenacin had fewer and less diverse communities of bacteria when evaluated by PCR and extended urine cultures.

The clinical significance of the bacteria identified is not well understood. However, these studies show that the presence of bacteria is being missed by standard cultures. Dune et al. found that of patients with UTI symptoms, 27.5% were standard culture negative but extended quantitative urine culture positive. This demonstrates that practitioners may be overlooking urinary tract infections in patients with frequency and urgency. Therefore, if bacteria within the urine can be detected with extended cultures, can this technique be used to improve detection and treatment of urinary infections in patients with symptoms of frequency and urgency?

The hypotheses states that extended urine cultures are more sensitive in the identification of urinary tract infections in patients with symptoms of urgency and frequency. The secondary hypothesis is that treatment of the uropathogen identified on extended urine cultures will improve patient symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18 y/o-70 y/o
* Able to consent
* Urgency /Frequency
* Urge incontinence
* PUF score ≤ 4
* Bother questionnaire #2 or #3 answered either "a moderate amount" or "a lot"

Exclusion Criteria:

* Pregnant
* Pelvic radiation
* Chronic pelvic pain
* Urinary retention
* Greater than Stage 2 prolapse
* Renal calculi
* Recurrent UTI (2 in 6 months)
* Immunosuppressed
* Neurologic disorder
* No antibiotics in the past 4 weeks

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included in the study if they have a history of overactive bladder or urgency and frequency with or without incontinence, they must be female, able to speak English, and must be 18 years old or older and able to provide informed consent. Patients must have a PUF score of less than or equal to 4 and answer "a moderate amount" or "a lot" on the Bother questionnaire number 2 or 3. They must also not be a prisoner. Patients will be excluded if they have are pregnant, have urinary retention, greater than stage 2 prolapse, renal calculi, immune-suppressed, those with neurologic disorders, prior use of antibiotics in the past month, had prior radiation to the pelvic floor, or chronic pelvic pain defined by more than 6 months of pelvic pain, or dysuria.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of extended urine cultures compared to standard urine cultures. | one year
  Extended urine cultures are more sensitive in the identification of urinary tract infections in patients with symptoms of urgency and frequency then standard cultures as measured by a positive urine extended culture.

SECONDARY OUTCOMES:
Treatment of uropathogens found on extended cultures result in negative repeat extended urine culture. | one year
  Treatment of uropathogens found on extended cultures result in negative repeat extended urine culture.
Treatment of uropathogens found on extended cultures improves urinary tract symptoms measured by the Bother and UDI-6 questionnaires | one year
  Treatment of the uropathogen identified on extended urine cultures improve patient's urgency and frequency symptoms measured by the Bother and UDI-6 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hurtado, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Patient information will not be shared with outside researchers.

REFERENCES:
- [Background] Hilt EE, McKinley K, Pearce MM, Rosenfeld AB, Zilliox MJ, Mueller ER, Brubaker L, Gai X, Wolfe AJ, Schreckenberger PC. Urine is not sterile: use of enhanced urine culture techniques to detect resident bacterial flora in the adult female bladder. J Clin Microbiol. 2014 Mar;52(3):871-6. doi: 10.1128/JCM.02876-13. Epub 2013 Dec 26. PMID 24371246
- [Background] Pearce MM, Hilt EE, Rosenfeld AB, Zilliox MJ, Thomas-White K, Fok C, Kliethermes S, Schreckenberger PC, Brubaker L, Gai X, Wolfe AJ. The female urinary microbiome: a comparison of women with and without urgency urinary incontinence. mBio. 2014 Jul 8;5(4):e01283-14. doi: 10.1128/mBio.01283-14. PMID 25006228
- [Background] Thomas-White KJ, Hilt EE, Fok C, Pearce MM, Mueller ER, Kliethermes S, Jacobs K, Zilliox MJ, Brincat C, Price TK, Kuffel G, Schreckenberger P, Gai X, Brubaker L, Wolfe AJ. Incontinence medication response relates to the female urinary microbiota. Int Urogynecol J. 2016 May;27(5):723-33. doi: 10.1007/s00192-015-2847-x. Epub 2015 Sep 30. PMID 26423260
- [Background] Tanaka Dune, Evann Hilt, Travis Price, Colleen Fitzgerald, Cynthia Brincat, Linda Brubaker, Alan J. Wolfe, Paul Schreckenberger, Elizabeth R. Mueller. False negatives of standard urine cultures may delay patient treatment. AUGS. October 13-17, 2015.